CLINICAL TRIAL: NCT03571828
Title: A Phase 1, First-in-Human, Open-Label Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of AMG 562 in Subjects With Relapsed / Refractory Diffuse Large B-cell Lymphoma, Mantle Cell Lymphoma, or Follicular Lymphoma
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of AMG 562 in Subjects With r/r Diffuse Large B-cell Lymphoma, Mantle Cell Lymphoma, or Follicular Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Amgen decided to discontinue study because of a business decision and not because of safety reasons
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20170533
Record Dates: First submitted 2018-06-18; First posted 2018-06-28 (Actual); Results first posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2023-09

CONDITIONS: Diffuse Large B-cell Lymphoma(DLBCL); Mantle Cell Lymphoma (MCL); Follicular Lymphoma (FL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Exploration (Experimental): Dose exploration cohorts to estimate the MTD, safety, tolerability, and PK of different doses of AMG 562 in subjects with relapsed/refractory DLBCL, MCL or FL using a Bayesian logistic regression model (BLRM; Neuenschwander et al, 2008).
  Interventions: Drug: AMG 562
- Part 2: Dose Expansion (Experimental): dose expansion part to gain further clinical experience, safety and efficacy data for AMG 562 in subjects with relapsed / refractory DLBCL. The dose to be evaluated will be at or below the MTD estimated in the dose exploration cohorts.
  Interventions: Drug: AMG 562

INTERVENTIONS:
Drug: AMG 562 — AMG 562 is a BiTE® antibody construct that targets CD19 and is intended for the treatment of patients with B-cell malignancies.

SUMMARY:
Evaluate the safety and tolerability of AMG 562 in adult subjects with DLBCL, MCL, or FL. Estimate the maximum tolerated dose (MTD) and/or a biologically active dose (e.g., recommended phase 2 dose [RP2D])

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study-specific activities/procedures
* Age ≥ 18 at the time of informed consent.
* Biopsy proven B-NHL including:

  * DLBCL, which also includes DLBCL that represents transformation of indolent NHL (including follicular, marginal zone, and lymphoplasmacytic lymphoma excluding chronic lymphocytic leukemia or Hodgkin Lymphoma) and DLBCL with alterations of MYC and BCL2 and/or BCL6 also described as double-hit and triple-hit lymphomas.
  * FL
  * MCL Presentations of these histologies with substantial occurrence of malignant cells into the bloodstream (lymphocyte count ≥ 7 x 10^9/L) including all leukemic presentations are excluded.

The following histologies are not eligible:

Lymphoblastic lymphoma Burkitt lymphoma Any histologies not specifically mentioned must be discussed with the Medical Monitor

* Subjects with transformation of indolent lymphoma must have received therapy after a diagnosis of transformation that is appropriate for aggressive histology.

  - Subjects who received prior CD19-targeting treatment are allowed (CAR-T cell therapy is excluded). A biopsy following CD19-targeting treatment is required unless no lesions are accessible or the risk of the biopsy is deemed too high by the investigator For Part 2 (Expansion in patients with DLBCL): only biopsy proven DLBCL (biopsy proven at least at primary diagnosis), including DLBCL that represents transformation of indolent NHL (including follicular, marginal zone, and lymphoplasmacytic lymphoma excluding chronic lymphocytic leukemia or Hodgkin Lymphoma) are eligible. Other histologies are not eligible.
* Presentations of these histologies with substantial occurrence of malignant cells into the bloodstream (lymphocyte count ≥ 7 x 10^9/L) including all leukemic presentations are excluded.
* Subjects with transformation of indolent lymphoma must have received therapy after a diagnosis of transformation that is appropriate for aggressive histology as described in inclusion criterial.
* Subjects who received prior CD19-targeting treatment are allowed (CAR-T cell therapy is excluded) A biopsy following CD19-targeting treatment is required unless no lesions are accessible or the risk of the biopsy is deemed too high by the investigator - For DLBCL: Refractory (no prior CR/CMR) to first or later line of treatment or relapsed (prior CR/CMR) after two or more prior treatments, with at least one treatment consisting of standard multiagent chemotherapy containing an anthracycline AND an approved anti-CD20 agent. Examples of appropriate therapy include but are not limited to R-CHOP (14 or 21), R-CHOEP, and DA-R-EOCH.

For FL: Refractory (no prior CR/CMR) to first or later line of treatment or relapsed (prior CR/CMR) after three or more prior treatments, with at least one treatment consisting of a standard chemotherapy containing an approved anti-CD20 agent.

Examples of appropriate therapy include but are not limited to R-CHOP, R-CVP, and BR.

For MCL: Refractory (no prior CR/CMR) to first or later line of treatment or relapsed (prior CR/CMR) after three or more prior treatments, with at least one treatment consisting of a standard chemotherapy containing an approved anti-CD20 agent. Examples of appropriate therapy include but are not limited to R-CHOP, BR and hyper-CVAD alternating with R-MTX/Ara-C.

For subjects with refractory B-NHL and who have received radiotherapy, PET positivity should be demonstrated no less than 6 weeks after the last dose of radiotherapy

* Minimum life expectancy of 12 weeks
* Radiographically measurable disease with a clearly demarcated nodal lesion at least 1.5 cm in its largest dimension or a target extranodal lesion at least 1.0 cm in its largest dimension. In the dose exploration phase in case disease is not radiographically measurable PET positivity (ie, Deauville ≥4) instead is acceptable.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Laboratory parameters (completed within 14 days prior to enrollment):

Hematology:

* Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L
* Platelets ≥ 75 x 10^9/L

Chemistry:

* Creatinine clearance ≥ 60 mL/min (calculated using Cockcroft Gault equation)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 3X upper limit of normal (ULN)
* Total bilirubin (TBL) < 2x ULN (unless Gilbert's disease or if liver involvementwith lymphoma)

Exclusion Criteria:

* Treatment within 30 days prior to enrollment with another investigational device or drug (interventional clinical study / studies). Other investigational procedures while participating in this study are excluded (observational studies are permitted).
* Prior anti-cancer therapy as specified below:

  * At least 6 weeks must have elapsed since any prior systemic inhibitory/stimulatory immune checkpoint molecule therapy (eg, ipilimumab, nivolumab, pembrolizumab, atezolizumab, OX40 agonists, 4-1BB agonists, etc) before the first dose of AMG 562.
  * Other targeted anti-cancer therapy (chemotherapy, molecular targeted therapy, steroids) within 14 days or 5 half lives (which ever is longer) prior to first dose of AMG 562. Patients requiring continued treatment due to aggressive disease may only be included if there is agreement by both the investigator and the Amgen Medical Monitor.
  * Radiation therapy completed within 28 days prior to first dose of AMG 562.
  * Autologous HSCT within six weeks prior to start of AMG 562 treatment.
  * At least 4 weeks must have elapsed since any prior treatment with antibody therapy (exception immune checkpoint inhibitors) before the first dose of AMG 562.
* Prior CD19-directed CAR-T cell therapies
* Prior allogeneic HSCT.
* For Part 2 (Expansion in patients with DLBCL): fluorodeoxyglucose non-avid patients.
* Baseline electrocardiogram (ECG) QTc > 470 msec.
* Autoimmune disorders requiring chronic systemic steroid therapy or any other form of immunosuppressive therapy. Patient may be included if the treatment is discontinued more than 3 months prior to the first dose of AMG 562 at a low likelihood of relapse AND if there is agreement by both the investigator and the Amgen Medical Monitor.
* Unresolved toxicity from prior anti-tumor therapy, defined as not having resolved to CTCAE version 4.0 grade 1, or to levels dictated in the eligibility criteria with the exception of alopecia or toxicities from prior anti-tumor therapy that are considered irreversible (defined as having been present and stable for > 28 days) which may be allowed if they are not otherwise described in the exclusion criteria AND there is agreement to allow by both the investigator and the Amgen Medical Monitor.
* Presence of clinically relevant central nervous system (CNS) pathology such as epilepsy, paresis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis.
* Evidence of CNS involvement by NHL.
* Known infection with human immunodeficiency virus (HIV).
* Exclusion of hepatitis infection based on the following results and/or criteria:

  * Positive for hepatitis B surface antigen (HBsAg) (indicative of chronic hepatitis B or recent acute hepatitis B).
  * Negative HBsAg and positive for hepatitis B core antibody: Assay for hepatitis B virus DNA by polymerase chain reaction (PCR) is necessary. Detectable hepatitis B virus DNA suggests occult hepatitis B.
  * Positive Hepatitis C virus antibody (HCVAb): Assay for hepatitis C virus RNA by PCR is necessary. Detectable hepatitis C virus RNA suggests chronic hepatitis C.
* History of malignancy other than B-NHL within the past 3 years with the exception of:

  * Malignancy treated with curative intent and with no known active disease present for ≥ 3 years before enrollment and felt to be at low risk for recurrence by the treating physician.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated cervical carcinoma in situ without evidence of disease.
  * Adequately treated breast ductal carcinoma in situ without evidence of disease.
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer.
  * Adequately treated urothelial papillary noninvasive carcinoma or carcinoma in situ.
* Major surgery within 28 days of first dose AMG 562.
* History of arterial thrombosis (eg, stroke or transient ischemic attack) within 12 months of first dose of AMG 562.
* Presence of fungal, bacterial, viral, or other infection requiring IV antimicrobials for management within 7 days of first dose AMG 562. NOTE: Simple UTI and uncomplicated bacterial pharyngitis are permitted after consultation with sponsor and if responding to active treatment.
* Subject has known sensitivity to immunoglobulins or any of the products or components to be administered during dosing.
* Males and females of reproductive potential who are unwilling to practice highly effective method(s) of birth control while on study through 110 days (females) and 170 days (males) after receiving the last dose of study drug. Highly effective methods of birth control include sexual abstinence (males, females); vasectomy; bilateral tubal ligation/occlusion; or a condom with spermicide (males) in combination with hormonal birth control or intrauterine device (IUD) (females).
* Females who are lactating/breastfeeding or who plan to breastfeed while on study through 110 days after receiving the last dose of study drug.
* Females with a positive pregnancy test.
* Females planning to become pregnant while on study through 110 days after receiving the last dose of study drug.
* Males who are unwilling to abstain from sperm donation while on study through 170 days after receiving the last dose of study drug.
* Subjects likely to not be available to complete all protocol- required study visits or procedures including BM aspirates/biopsies, and/or to comply with all required study procedures to the best of the subject and investigator's knowledge.
* History or evidence of any other clinically-relevant concurrent disorder, condition or disease (eg, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia requiring therapy at time of screening) with the exception of those outlined above that, in the opinion of the investigator or Amgen medical monitor, if consulted, would not pose a risk to subject safety or interfere with the study evaluation, procedures or completion.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (12):
- United States (7):
  - City of Hope National Medical Center, Duarte, California
  - University of California Los Angeles, Los Angeles, California
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
- Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven, Belgium
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Germany (3):
  - Klinikum der UniversitÃ¤t MÃ¼nchen Campus GroÃŸhadern, MÃ¼nchen
  - Universitatsklinikum Ulm, Ulm
  - UniversitÃ¤tsklinikum WÃ¼rzburg, WÃ¼rzburg

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 13 centers in United States, Canada, South Korea, Germany, and Japan from October 2018 to January 2022.
Pre-assignment Details: The study planned to consist of 2 parts. Part 1 included a dose exploration and Part 2 a dose-expansion group. However, no participants were enrolled into Part 2.
Groups:
- Cohort 1: AMG 562 0.1 μg: Participants with relapsed/refractory diffuse large B-cell lymphoma (DLBCL), mantle cell lymphoma (MCL), or follicular lymphoma (FL) received AMG 562 0.1 μg administered as once weekly intravenous (IV) infusions for up to approximately 8 months.
- Cohort 2: AMG 562 0.3 μg: Participants with relapsed/refractory DLBCL, MCL, or FL received AMG 562 0.3 μg administered as once weekly IV infusions for up to approximately 8 months.
Period: Overall Study
Arm/Group | Cohort 1: AMG 562 0.1 μg | Cohort 2: AMG 562 0.3 μg
Started | 9 | 1
Received Investigational Product | 8 | 1
Completed | 1 | 0
Not Completed | 8 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Decision by sponsor | 5 | 1
Not completed — Death | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All participants who received at least one dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: AMG 562 0.1 μg | Cohort 2: AMG 562 0.3 μg | Total
Number analyzed (Participants) | 8 | 1 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (6.8) | 66.0 (NA) — Standard deviation (SD) could not be calculated as Cohort 2 only included 1 participant. | 63.6 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 1 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 1 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose Limiting Toxicity (DLT)
Time Frame: Day 1 to Day 28
Population: DLT Analysis Set: all participants who either experienced DLTs or completed 28 days of DLT observational period and did not experience DLTs.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: AMG 562 0.1 μg | Cohort 2: AMG 562 0.3 μg
Number analyzed (Participants) | 6 | 1
Participants | 1 | 0

2. Primary Outcome: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical trial participant. TEAEs were any AE that occurred after receiving at least 1 dose of treatment.
  Treatment-related TEAEs were those considered related to study treatment by the investigator.
  Disease-Related TEAEs were events (serious or non-serious) anticipated to occur in the study population due to the underlying disease.
  Any clinically significant changes in vital signs, physical examinations, electrocardiograms (ECG)s and clinical laboratory tests were recorded as TEAEs.
Time Frame: Up to 2 years
Population: Safety Analysis Set: All participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: AMG 562 0.1 µg: Participants with relapsed/refractory diffuse large B-cell lymphoma (DLBCL), mantle cell lymphoma (MCL), or follicular lymphoma (FL) received AMG 562 0.1 μg administered as once weekly intravenous (IV) infusions for up to approximately 8 months.
Arm/Group | Cohort 1: AMG 562 0.1 µg | Cohort 2: AMG 562 0.3 μg
Number analyzed (Participants) | 8 | 1
Participants
  TEAEs | 8 | 1
  Treatment-related TEAEs | 4 | 0
  Disease-related TEAEs | 1 | 0

3. Secondary Outcome: Maximum Observed Concentration (Cmax) of AMG 562
Time Frame: Day 1
Population: Pharmacokinetic (PK) Analysis Set: all participants who have received at least 1 dose of AMG 562 and have at least 1 PK sample collected.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: AMG 562 0.1 µg | Cohort 2: AMG 562 0.3 μg
Number analyzed (Participants) | 4 | 0
ng/mL | 0.0460 (0.0173) |

4. Secondary Outcome: Time of Maximum Concentration (Tmax) of AMG 562
Time Frame: Day 1
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: AMG 562 0.1 µg | Cohort 2: AMG 562 0.3 μg
Number analyzed (Participants) | 4 | 0
hours | 1.2 [1.0 to 6.1] |

5. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Timepoint (AUClast) of AMG 562
Time Frame: Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cohort 1: AMG 562 0.1 µg | Cohort 2: AMG 562 0.3 μg
Number analyzed (Participants) | 3 | 0
hr*ng/mL | 0.658 (0.426) |

6. Secondary Outcome: Half-life (t1/2) of AMG 562
Time Frame: Day 22
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: AMG 562 0.1 µg | Cohort 2: AMG 562 0.3 μg
Number analyzed (Participants) | 1 | 0
hours | 61.2 [NA to NA] — Only 1 participant had evaluable data, so lower and upper limit could not be calculated. |

7. Secondary Outcome: Objective Response Rate (ORR) Per Lugano Classification
Description: ORR was defined as the percentage of participants with a confirmed complete metabolic response (CMR) or partial metabolic response (PMR) as defined by Lugano Classification.
  Per the Lugano Classification, positron emission tomography-computed tomography (PET-CT) were defined on the 5-point scale as scores 1, 2, or 3 (where 1 = no uptake above background; 2 = uptake </= mediastinum; and 3 = uptake > mediastinum but </= liver) and PET-positive scans, as scores of 4 or 5 (where 4 = uptake moderately higher than liver; 5 = uptake markedly higher than liver and/or new lesions).
  CMR: score of 1, 2 or 3 in nodal or extranodal sites with or without a residual mass.
  PMR: score of 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size.
Time Frame: Day 1 up to 2 years
Population: Safety Analysis Set: All participants who received at least one dose of investigational product.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: AMG 562 0.1 µg | Cohort 2: AMG 562 0.3 μg
Number analyzed (Participants) | 8 | 1
Percentage of participants
  CMR | 12.5 | 0.0
  PMR | 0.0 | 0.0

8. Secondary Outcome: Best Overall Response Per Lugano Classification
Description: Per the Lugano Classification, positron emission tomography-computed tomography (PET-CT) were defined on the 5-point scale as scores 1, 2, or 3 (where 1 = no uptake above background; 2 = uptake </= mediastinum; and 3 = uptake > mediastinum but </= liver) and PET-positive scans, as scores of 4 or 5 (where 4 = uptake moderately higher than liver; 5 = uptake markedly higher than liver and/or new lesions).
  CMR: score of 1, 2 or 3 in nodal or extranodal sites with or without a residual mass.
  PMR: score of 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size.
  No metabolic response (NMR): score of 4 or 5 with no obvious change in fluorodeoxyglucose (FDG) uptake.
  Progressive metabolic disease (PMD): score 4 or 5 in any lesion with an increase in intensity of FDG uptake from baseline (and/or new FDG-avid foci consistent with lymphoma).
Time Frame: Day 1 up to 2 years
Population: Safety Analysis Set: All participants who received at least one dose of investigational product.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: AMG 562 0.1 µg | Cohort 2: AMG 562 0.3 μg
Number analyzed (Participants) | 8 | 1
Percentage of participants
  CMR | 12.5 | 0.0
  PMR | 0.0 | 0.0
  NMR | 0.0 | 0.0
  PMD | 50.0 | 100.0
  Unable to Evaluate or Not Available | 37.5 | 0.0

9. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the date of an initial objective response per Lugano classification to the earlier of progression or death. Participants who had not ended their response at the time of analysis had DOR censored at their last disease assessment date.
Time Frame: Day 1 up to 2 years
Population: Safety Analysis Set - Objective Responders: All participants who received at least one dose of investigational product and had a CMR or PMR.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cohort 1: AMG 562 0.1 µg | Cohort 2: AMG 562 0.3 μg
Number analyzed (Participants) | 1 | 0
Days | NA (NA) — One participant in cohort 1 was censored and had completed study without disease progression or death, so DOR could not be calculated. |

10. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the interval from Day 1 to the earlier of a lymphoma progression or death from any cause; otherwise, PFS was censored at the last radiographic assessment date. If a participant had no post baseline radiographic assessment and a vital status of alive or unknown, PFS was censored at Day 1.
Time Frame: Day 1 up to 2 years
Population: Safety Analysis Set: All participants who received at least one dose of investigational product.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1: AMG 562 0.1 µg | Cohort 2: AMG 562 0.3 μg
Number analyzed (Participants) | 8 | 1
Months | 0.9 [0.6 to 8.1] | 1.0 [1.0 to 1.0]

11. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of Day 1 until death due to any cause. Any participant not known to have died at the time of analysis was censored based on the last recorded date on which the participant was alive.
Time Frame: Day 1 up to 2 years
Population: Safety Analysis Set: All participants who received at least one dose of investigational product.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Cohort 1: AMG 562 0.1 µg | Cohort 2: AMG 562 0.3 μg
Number analyzed (Participants) | 8 | 1
Months | NA [1.7 to NA] — Not enough participants experienced an event of death, so OS or the upper limit could not be calculated. | NA [NA to NA] — Not enough participants experienced an event of death, so OS could not be calculated.

ADVERSE EVENTS:
Time Frame: Mortality: Day 1 up to end of study, median time on study was 3.14 months (min: 0.30; max: 22.97) Adverse events: Day 1 up to 30 days after last dose, median time was 1.71 months (min: 1.35; max 22.64)
Description: Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug. Mortality reporting is reported for all participants enrolled.
Arm/Group | Cohort 1: AMG 562 0.1 μg | Cohort 2: AMG 562 0.3 μg
All-Cause Mortality (participants affected / at risk) | 2/9 | 0/1
Serious Adverse Events (participants affected / at risk) | 3/8 | 1/1
Other Adverse Events (participants affected / at risk) | 8/8 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: AMG 562 0.1 μg (N=8) | Cohort 2: AMG 562 0.3 μg (N=1)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: AMG 562 0.1 μg (N=8) | Cohort 2: AMG 562 0.3 μg (N=1)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Oesophageal pain (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 0
Pyrexia (General disorders) | 5 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Blood cholesterol increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0
Serum ferritin increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Non-Hodgkin's lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Areflexia (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Hypotonia (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Nephropathy (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
Amgen decided not to continue development of AMG 562 because of a business decision and not because of safety reasons. No conclusions can be drawn due to the small sample size of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT03571828/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT03571828/SAP_001.pdf